CLINICAL TRIAL: NCT06297213
Title: A Single and Repeat Dosing Study of the Safety, Drug Exposure and Clinical Activity of R-2487 in Patients With Sjogren's Syndrome (SS)
Brief Title: R-2487 in Patients With Sjogren's Syndrome (SS)
Acronym: R-2487-SS-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2487-SS-01
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Sjogren's Syndrome; Sjögren; Sjögren Syndrome, Unspecified
Keywords: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Other): Probiotic
  Interventions: Drug: R-2487

INTERVENTIONS:
Drug: R-2487 — R-2487 DP
  Other Names: Probiotic

SUMMARY:
The goal of this study is to determine the safety and tolerability of orally taken probiotic (R-2487) in patients with Sjogren's Syndrome.

Patients will take an oral dosage of probiotic (R-2487) and physicians will assess and measure their Sjogren's Syndrome. Blood and fecal evaluations of inflammation and assessment of probiotic (R-2487) on fecal level will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SS according to American-European Consensus Group Criteria
* Able to provide informed consent
* Subjects receiving prednisone (10 mg or less/day) must be on a stable dose for more than 2 weeks
* All male and female subjects who are biologically capable of having children must agree to use medically acceptable method of birth control for the duration of the study. All female subjects who are biologically capable of having children must have a negative pregnancy test result before administration of investigational product.
* The use of probiotics prior to study enrollment is accepted; however, during the course of the study, the use of probiotics is forbidden.

Exclusion Criteria:

* No known active overlapping or associated other autoimmune disease
* Prior allogenic or autologous bone marrow or organ transplantation
* Subjects with prior irradiation to the head and neck, including radioactive iodine treatment for hyperthyroidism
* Subjects who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Subjects who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations.
* Subjects with positive results for human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Subjects with active viral, bacterial, or fungal infection, or history of severe opportunistic infection within the preceding 3 months, or COVID-19 infection in the past 3 months
* Subjects with evidence of active or latent tuberculosis
* Active infection of the salivary or lacrimal glands
* Prior immunotherapy, biologics, or investigational therapy must have completed at least 5 half-lives or 30 days, whichever is longer, prior to the first dose of R-2487 DP
* Pregnant or breastfeeding women
* Current clinical findings of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, endocrine, neurological, or cerebral disease with laboratory values as following:

Hemoglobin level < 9.0 g/dL

Absolute white blood cell (WBC) count of <3.0×109/L (<3000/mm3), or absolute neutrophil count of <1.2×109/L (<1200/mm3), or absolute lymphocyte count of <0.8×109/L (<800/mm3).

Thrombocytopenia, defined by platelet count <100×109/L (<100,000/mm3)

Chronic kidney disease defined as Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, based on the age appropriate calculation.

Proteinuria ≥3+.

Total bilirubin (T-bili), aspartate aminotransferase (AST), alanine aminotransferase (ALT) more than 1.5 times upper limit of normal (ULN).

Previously diagnosed hepatic cirrhosis (Child Pugh A or higher) or previously diagnosed significant liver fibrosis (> F3)

* Any form of vaccination in the last 30 days, to include but not limited to influenza, COVID, shingles, tetanus, hepatitis, pneumonia, HPV, DPT, MMR, and polio.
* Subjects should not receive any of the following medications:

Rituximab or belimumab within 6 months prior to Day 1 Abatacept within 3 months prior to Day 1 Infliximab, Adalimumab, Certolizumab, Tocilizumab, Cyclosporine, or Mycophenolate mofetil within 2 months prior to Day 1 Etanercept, Anakinra, Immunoglobulin, or blood products within 28 days prior to Day 1

* Prior immunotherapy, including systemic corticosteroids, such prednisone, biologics, Janus kinase (JAK) inhibitors (such as tofacitinib, or upadacitinib), ozanimod, or investigational therapy must have completed at least 5 half-lives or 30 days, whichever is longer, prior to Day 0, unless otherwise specified. In the case of cell-depleting therapies, such as B or T cell depletion, cell counts must have recovered to acceptable or baseline levels (use of licensed agents for indications not listed in the package insert is permitted).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and their relationship to R-2487 (probiotic) administration | Baseline through Week 4
  To assess the number of participants with treatment-related adverse events after taking R-2487 (probiotic)

SECONDARY OUTCOMES:
Change in disease activity through Clinical European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ClinESSDAI) | Baseline through Week 4
  Change from Baseline in Disease Activity Score at Week 4 to assess the disease severity of Sjogren's syndrome using data without laboratory results
Change in Patient reported general health questionnaire Short Form Health Survey-36(SF-36) | Baseline through week 4
  Baseline Short Form Health Survey-36 (SF-36) Score over time. The Baseline Short Form Health Survey is the numerical sum of 36 patient reported outcome parameters of quality of life. The higher the score the more favorable the reflection of the quality of life.